CLINICAL TRIAL: NCT00877513
Title: Insulin Resistance in Smokers Undergoing Smoking Cessation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding expired
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-02-2165
Record Dates: First submitted 2009-02-23; First posted 2009-04-07 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Disease; Insulin Resistance
Keywords: Smoking; Insulin resistance; Metabolic syndrome; Body fat distribution; Cigarette smoking
MeSH Terms: conditions — Cardiovascular Diseases; Insulin Resistance; Smoking; Metabolic Syndrome; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Smokers (Experimental): Cigarette smokers wishing to quit
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Smoking cessation — Smoking cessation program over 8 weeks, consisting of cognitive behavioral counseling every 2 weeks along with adjunctive use of bupropion

SUMMARY:
Cigarette smoking increases CVD risk and worsens insulin resistance, but also contributes to weight loss; smoking cessation reduces CVD risk and improves insulin sensitivity, but also contributes to weight gain. The mechanisms that underlie these metabolic changes of cigarette smoking and smoking cessation on insulin resistance, body composition, and fat distribution are poorly understood.

DETAILED DESCRIPTION:
This study is a prospective, open cohort study of smokers who undergo a smoking cessation program, and who subsequently may or may not resume smoking spontaneously. Eligible subjects will be characterized at baseline with respect to their metabolic and CVD risk profiles, body fat composition and distribution. Subjects will then undergo an intensive 8-week smoking cessation program using bupropion plus cognitive behavioral counseling. Those who successfully abstain will be reassessed. Since most individuals who quit smoking will naturally resume smoking again over time, subjects will be assessed again after an additional 4 months of follow-up when a subset of subjects will be expected to have naturally resumed smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 70 inclusive; any ethnicity
* Cigarette smoking for at least 3 years, at a rate of at least 1 but not more than 2 packs per day
* BMI 19 kg/m2 or greater and 40 kg/m2 or less
* Willing to enter, and be able to comply with the instructions and scheduled follow-up of a smoking cessation program

Exclusion Criteria:

* Any physical disabilities that prevent the subject from participating in the study, as determined by the investigators
* History of CVD (ventricular arrhythmias, atrial arrhythmias with a history of hemodynamic instability, unstable angina, myocardial infarction, invasive coronary revascularization, or any hospitalization for CVD within the last 3 years, NYHA Class III or IV CHF)
* Current abuse of illicit drugs or heavy ethanol use
* History or baseline laboratory evidence of diabetes mellitus
* History of chronic obstructive pulmonary disease (COPD)
* BMI < 19 or > 40 kg/m2
* Subjects not following a regular diet and lifestyle pattern (e.g, homeless)
* Uncontrolled hypertension (BP 170 mmHg or greater systolic or 110 mmHg or greater diastolic)
* Fasting triglycerides 700 mg/dL or greater, or LDL-cholesterol 200 mg/dL or greater
* History of chronic renal or liver disease (hepatic transaminase elevations > 3 times the upper limit of the normal range; creatinine > 1.5 mg/L), malignancies not currently in remission, gastrointestinal disorders that interfere with nutrition; history of malnutrition, chronic infections (including HIV), or recent (within 30 days) surgeries or hospitalizations
* Concurrent use of medications that may alter metabolic parameters (including metformin, sulfonylurea agents, thiazolidinediones, weight loss agents, androgens or systemic glucocorticoids); lipid-lowering agents and oral contraceptives will be permitted as long as formulations, dosages and adherence remain unchanged throughout the course of the study. Oral contraceptives that are started during the course of the study will require the subject to be withdrawn from the study
* Perimenopausal women experiencing irregular menses, because of changing metabolic status during the perimenopause; these patients may be included if menses have ceased for at least 6 months
* Women who are pregnant, seeking to become pregnant in the next 6 months, or who are breastfeeding
* Any history of depression, suicidality, or any contraindications to bupropion (history of seizures, anorexia or bulimia)
* Current use of nicotine replacement products (gum or patch)
* Any other factors that, in the opinion of the investigators, may interfere with the safe conduct, successful completion, or data integrity of the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity by euglycemic hyperinsulinemic clamp | 8 weeks, 6 months

SECONDARY OUTCOMES:
Body mass index | 8 weeks, 4 months, 6 months
Body composition | 8 weeks, 4 months, 6 months
Body fat distribution | 8 weeks, 4 months, 6 months
Blood pressure | 8 weeks, 4 months, 6 months
Fasting lipid profile | 8 weeks, 4 months, 6 months
Apolipoproteins | 8 weeks, 4 months, 6 months
Fasting plasma glucose | 8 weeks, 4 months, 6 months
HOMA-IR index | 8 weeks, 4 months, 6 months
Adipokines | 8 weeks, 4 months, 6 months
Highly-sensitive C-reactive protein | 8 weeks, 4 months, 6 months
Morning cortisol | 8 weeeks, 4 months, 6 months
IGF-1 | 8 weeks, 4 months, 6 months
Mean total daily caloric intake | 8 weeks, 4 months, 6 months
Mean total daily caloric expenditure | 8 weeks, 4 months, 6 months
Suppression of hepatic glucose production by clamp | 8 weeks, 6 months
Resting energy expenditure by calorimetry | 8 weeks, 6 months
Oxidative and non-oxidative glucose disposal by clamp | 8 weeks, 6 months
Total energy expenditure under hyperinsulinemia by clamp | 8 weeks, 6 months
Fat oxidation under hyperinsulinemia by clamp | 8 weeks, 6 months
Fatty acid suppression under hyperinsulinemia by clamp | 8 weeks, 6 months
Adverse events | 8 weeks, 4 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States